CLINICAL TRIAL: NCT02922413
Title: Safety and Efficacy of Panhematin™ for Prevention of Acute Attacks of Porphyria
Brief Title: Panhematin for Prevention of Acute Attacks of Porphyria
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 14-0188; FD-R-03720 (Other Grant/Funding Number: FDA - OOPD)
Record Dates: First submitted 2016-01-01; First posted 2016-10-04 (Estimated); Results first posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Acute Intermittent Porphyria; Hereditary Coproporphyria; Variegate Porphyria
Keywords: Porphyria; Heme
MeSH Terms: conditions — Porphyria, Acute Intermittent; Coproporphyria, Hereditary; Porphyria, Variegate; Porphyrias | interventions — Hemin; Injections

STUDY DESIGN:
Intervention Model Description: Two group parallel blinded study comparing active drug and placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Administered doses are shielded from view. The pharmacy and one nurse who administers the drug intravenously will not be blinded.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hemin for injection (Experimental): Double blind doses of Panhematin 4 mg/kg body weight reconstituted with 25% human albumin and infused over at least one hour.
  Interventions: Biological: Hemin for injection
- Placebo (Placebo Comparator): A double blind dose of saline.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Hemin for injection — Panhematin 4 mg/kg body weight reconstituted with 25% human albumin infused intravenously over at least 1 hour.
  Other Names: Hematin
  Arms: Hemin for injection
Other: Placebo — Saline infusion
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if Panhematin is safe and effective for prevention of acute attacks of porphyria.

The study aims to provide high quality evidence for the use on hemin for prevention of acute attacks of porphyria. High quality studies have not been done previously for treating or preventing acute attacks with hemin. The lack of strong evidence for efficacy of hemin for treatment and prevention of attacks limits its availability for patients with acute porphyrias. Funding source: FDA Office of Orphan Product Development (FDA OOPD) FD-R-03720

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled, parallel group trial investigating the efficacy and safety of Panhematin™ for preventing acute attacks in at least 20 subjects with well-documented acute porphyria (acute intermittent porphyria, hereditary coproporphyria or variegate porphyria). Subjects will (1.) have had frequent attacks in the past, with symptoms such as abdominal, back and/or limb pain and diagnosed after exclusion of other causes, and (2.) be on hemin prophylaxis for prevention of frequent attacks. It is expected that they will have had 6 or more attacks in one year before starting hemin prophylaxis. This would be considered justification for a preventive regimen of hemin on clinical grounds. Double blind Panhematin™ or placebo will be given. The number of doses will correspond to the number of doses that a subject receives in approximately one week for their prophylactic regimen. An interim analysis will be carried out after completion of 10 subjects to assess progress and possibly adjust the sample size. The trial consists of the following visits:

* A screening visit to determine eligibility and obtain informed consent.
* A treatment visit for administration of double blind prophylactic doses of Panhematin™ or placebo corresponding to the number of doses the subject receives for their prophylactic regimen within approximately one week.
* Follow up visit at 1, 2, 3, and 4 weeks to assess response to the infusion of Panhematin™ or placebo. These visits will be in person or by telephone.
* Additional visits may be scheduled if needed, for example for treatment of symptoms.
* Follow-up visits 3 and 6 months after the end of treatment either in person or by telephone Subjects will have laboratory documentation of one of the acute porphyrias. Molecular documentation is also expected, although rarely a causative mutation cannot be detected. Upon entry into the study they will be given in a blinded fashion one or more preventive doses of either Panhematin™ (4 mg/kg) or placebo, the number of which will correspond to the number of prophylactic doses they have been receiving within approximately one week for prophylaxis. A recurrent attack within the next 1, 2, 3 and 4 weeks will represent treatment failures. Because at study entry most subjects are expected to be on weekly prophylactic hemin treatment, and hemin is a short-acting drug, emphasis in the analysis will be on attacks occurring within 1 week after study treatment.

Any attacks that occur during the study will be treated according to standard of care, which may include Panhematin™, either at the study site or at a subject's usual treatment location.

It is intended that 20 subjects will complete treatment with blinded treatment and at least 4 weeks of follow up. A completed subject is one who meets all entrance criteria, has no exclusion criteria and completes the single dosing and at least one week of follow up, or is withdrawn because of an adverse event.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 years
2. Willing to provide written informed consent
3. A diagnosis of acute intermittent porphyria, hereditary coproporphyria or variegate porphyria confirmed by the following criteria, which are based on the criteria for enrollment in the Longitudinal Study of the Porphyrias Consortium. For each type of porphyria, the inclusion criteria are based on 1) clinical features, 2) biochemical findings, as documented by laboratory reports (or copies) of porphyria-specific testing, and 3) molecular studies to identify a mutation in a porphyria-related gene. Equivocal biochemical measurements may require confirmatory testing. Testing for a disease-causing mutation must be attempted, but an identified mutation is not essential for enrollment, since it is known that a mutation cannot be found in a small fraction (<5%) of biochemically proven cases of porphyria. Subjects will (1.) have had frequent attacks in the past, with symptoms such as abdominal, back and/or limb pain and diagnosed after exclusion of other causes, and (2.) be on hemin prophylaxis for prevention of frequent attacks. It is expected that they will have had 6 or more attacks in one year before starting hemin prophylaxis.

Exclusion Criteria:

1. Symptoms such as abdominal, back or limb pain are explained by another condition, as judged by the investigator
2. Known or suspected allergy to Panhematin™ or related products
3. A known or suspected allergy to human albumin
4. Any disease or condition that the investigator judges would lead to an unacceptable risk to the patient or interfere with the successful collection of data for the trial
5. Previous randomization in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-10-30 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2023-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karl E Anderson, MD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hemin for Injection | Placebo
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hemin for Injection | Placebo | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 13
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 6 | 13
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Acute Attacks of Porphyria After Treatment
Description: Participants were interviewed weekly by telephone to record the number of acute porphyria attacks after initial treatment with Panhematin or placebo.
Time Frame: 1-4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Hemin for Injection | Placebo
Number analyzed (Participants) | 7 | 6
Participants | 1 | 5
Statistical Analysis 1: Comparison: Hemin for Injection vs Placebo; Test type: Superiority; p = 0.029, 2-sided Fisher's Exact Test

2. Primary Outcome: Number of Participants With Treatment-Related Serious Adverse Events
Description: The number of participants who experience treatment-related serious adverse events (SAEs) as assessed and graded using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Time Frame: 1-4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Hemin for Injection | Placebo
Number analyzed (Participants) | 7 | 6
Participants | 0 | 0

3. Other Pre Specified Outcome: Effects on Levels of Porphobilinogen
Description: To evaluate the biochemical effects of Panhematin™ in patients treated with Panhematin™ to prevent attacks of acute porphyria by measuring urinary porphobilinogen and serum porphobilinogen. This will determine whether biochemical measurements are predictive of efficacy in preventing an attack.
Time Frame: 1-4 weeks
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Effects of Age
Description: To evaluate effects of age, as an example of clinical features, on response to preventive administration of Panhematin™.
Time Frame: 1-4 weeks
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Effects of the Nature of the Porphobilinogen Deaminase (PBGD) Mutation
Description: To evaluate effects of the nature or the PBGD mutation on response to preventive Panhematin™
Time Frame: 1-4 weeks
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Frequency of Injection Site Complications
Description: To evaluate the use of Panhematin™ reconstituted with 25% human albumin in patients treated to prevent acute attacks of porphyria in terms of the frequency of injection site complications, which may include thrombosis or inflammation.
Time Frame: 1-4 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1-4 weeks
Arm/Group | Hemin for Injection | Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 0/7 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/13/NCT02922413/Prot_SAP_000.pdf